CLINICAL TRIAL: NCT03194321
Title: A Prospective, Pilot Trial to Evaluate Safety and Tolerability of Tacrolimus Extended-Release (Astagraf XL) in HLA Sensitized Kidney Transplant Recipients
Brief Title: Trial to Evaluate Safety and Tolerability of Tacrolimus Extended-Release (Astagraf XL) in Human Leukocyte Antigen (HLA) Sensitized Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Stanley Jordan, MD, Director, Nephrology & Transplant Immunology, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043132
Record Dates: First submitted 2017-05-24; First posted 2017-06-21 (Actual); Results first posted 2021-12-30 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: End Stage Renal Disease
Keywords: Highly-sensitized; Kidney transplantation; Desensitization
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tacrolimus Extended-Release Arm (Experimental): All patients will receive tacrolimus extended-release adjusted to target trough levels, mycophenolate mofetil or mycophenolate sodium, and prednisone per CSMC practice.
  Interventions: Drug: Tacrolimus Extended-Release Oral Capsule

INTERVENTIONS:
Drug: Tacrolimus Extended-Release Oral Capsule — Maintenance immunosuppression will consist of tacrolimus extended-release, mycophenolate mofetil 500mg twice daily or mycophenolate sodium 360mg twice daily, and prednisone.

SUMMARY:
The purpose of this study is to demonstrate the safety of tacrolimus extended-release in HLA sensitized (HS, defined as panel reactive antibody ≥ 30%), kidney transplant recipients after desensitization with intravenous immunoglobulin (IVIG) and rituximab (also known as ritux) +/- plasma exchange (PLEX) per the standard of care with alemtuzumab induction.

DETAILED DESCRIPTION:
The study will be a single center, pilot trial. It will be an open label, single-arm, non- controlled design. All HS kidney transplant recipients with Panel Reactive Antibodies (PRA) ≥ 30%, age 18 and older, requiring desensitization may be included in the study. Initial desensitization protocol for living donor (LD) or deceased donor (DD) includes Intravenous Immunoglobulin (IVIG) 2g/kg (>70kg max 140g) given on day 0 (split over 2 days for peritoneal dialysis patients), rituximab 375mg/m2 (rounded to the nearest 100mg vial) given on day 15, and IVIG 2g/kg (>70kg max 140g ) given on day 30. Recipients for LD or DD who are unresponsive to IVIG/ritux (after 2 months for LD and after 6 months for DD) will require PLEX 5-7 sessions followed by IVIG 2g/kg (>70kg max 140g) and rituximab 375mg/m2. Patients will be receiving acetaminophen, antihistamine, and steroid as premedication for all infusions.

A total of 20 subjects will be enrolled in the study. Subjects will take part in the study until they are one year post-transplant. All subjects will require informed consent. At the time of screening, subjects will receive a physical exam and undergo lab testing. Alemtuzumab 30mg, will be administered subcutaneously to all subjects for induction immunosuppression immediately post-transplant. Maintenance immunosuppression will consist of tacrolimus extended-release, mycophenolate mofetil 500mg twice daily or mycophenolate sodium 360mg twice daily, and prednisone. Patients will receive antimicrobial prophylaxis per Cedars-Sinai Medical Center (CSMC) protocol. Lab tests and physical exams for safety will take place according to the evaluation schedule below. Safety will be assessed by the reporting of serious adverse events.

Tacrolimus trough level, complete metabolic panel, liver function panel, complete blood count with differential, Donor Specific Antibodies (DSA), and urinalysis with culture will be assessed according to the evaluation schedule below. Subjects will complete the study at one year post-transplant. Consent may be withdrawn by the study participant at any time. The investigator may also withdraw the study participant at any time if there are any safety concerns.

Desensitization includes Intravenous Immunoglobulin (IVIG) 2g/kg (>70kg max 140g) given on day 0 (split over 2 days for peritoneal dialysis patients), rituximab 375mg/m2 (rounded to the nearest 100mg vial) given on day 15, and IVIG 2g/kg (>70kg max 140g ) given on day 30. Patients will require PLEX 5-7 sessions if they have received desensitization in the past. In this case, patients will receive PLEX daily x 5-7 sessions followed by IVIG 2g/kg (>70kg max 140g) and rituximab 375mg/m2. Patients will be receiving acetaminophen, antihistamine, and steroid as premedication for all infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of a deceased or living donor kidney allograft
2. Patients must have undergone desensitization with intravenous immunoglobulin (IVIG) and rituximab with or without plasma exchange prior to transplant or be administered IVIG and rituximab peri-operatively (within seven days of transplant) post-transplant
3. Age 18 and over
4. Able to understand and provide informed consent
5. Calculated Panel Reactive Antibodies (CPRA)> 30% demonstrated on 3 consecutive samples. The methodology to measure polymerase chain reaction (PCR) includes FLOW and Luminex Single Antigen Assay.
6. At transplant, patient must have an acceptable crossmatch (as defined as T-or B- Flow Cytometry Crossmatch (FCMX) ≤ 225 MCS) from non-HLA identical donor. Negative crossmatch is Tpronase FCMX <70; T- FCMX <50 and Bpronase FCMX <130; B-FCMX <100.

Exclusion Criteria:

1. Recipients of a dual simultaneous kidney/liver, kidney/heart, kidney/lung, or kidney/pancreas transplant
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
3. Patients being treated with drugs that are strong inducers or inhibitors of cytochrome P450 3A4
4. Patients with a clinically significant systemic infection within 30 days prior to transplant
5. Patients who have any surgical or medical condition that may affect absorption of drug, such as severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and/or excretion of study medication
6. Women of childbearing potential who are either pregnant, lactating, planning to become pregnant during this trial, or with a positive serum or urine pregnancy test. Women of childbearing potential must be willing to agree to contraceptive practices.
7. Patients who are PCR positive for Hep B, Hep C, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female HLA sensitized (HS) renal transplantation patients, 18 years of age and over, receiving a cadaveric or living donor kidney transplant may enter the study. Patients must receive desensitization therapy. Twenty patients will be enrolled at Cedars-Sinai Medical Center (CSMC) for this pilot study. Patients who discontinue the study prematurely will not be replaced.
Pre-assignment Details: Of the total 31 participants ages 18 years and older screened, 20 were enrolled in this single-center, open-label single-arm, non-controlled study.
Period: Overall Study
Arm/Group | Tacrolimus Extended-Release Arm
Started | 20
Completed | 17
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Travel for Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tacrolimus Extended-Release Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10.4956)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events and Treatment Failure
Description: To determine the safety of tacrolimus extended-release in HS kidney transplant recipients after desensitization with intravenous immunoglobulin (IVIG) and rituximab +/- plasma exchange (PLEX) per the standard of care and alemtuzumab induction. This will be measured by the rate of serious adverse events (SAEs) and treatment failure. Treatment failure is defined as a composite of biopsy proven acute rejection (BPAR), graft failure, or death. BPAR is defined as ≥ Banff 1A using the Banff 2007 criteria.
Time Frame: 12 months
Population: All participants who completed their 12 month visit were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus Extended-Release Arm
Number analyzed (Participants) | 17
Participants
  Active/Chronic Antibody Mediated Rejection (cABMR) | 2
  Chronic active Cell Mediated Rejection (CMR)/Antibody Mediated Rejection (ABMR) | 2
  Early Transplant Glomerulopathy (TG) | 1
  Cell Mediated Rejection (CMR) | 1
  Infections (i.e. BK Viremia, Cytomegalovirus (CMV))) | 4

2. Secondary Outcome: Change in Donor Specific Antibodies (DSA) as Defined by the DSA Relative Intensity Score (RIS)
Description: To observe the change in DSA as defined by the DSA RIS, which is defined by: 0 points for no DSA, 2 points for each weak DSA (MFI <5,000), 5 points for each moderate DSA (MFI 5,000 -10,000), and 10 points for each strong DSA (MFI >10,000).
Time Frame: Transplant, 1 month, 3 months, 6 months, 9 months, and 12 months
Population: All participants enrolled were assessed. Number of participants analyzed differed due to study withdrawals prior to 12 months.
Measure: Mean (Standard Deviation); unit: DSA Relative Intensity Score
Arm/Group | Tacrolimus Extended-Release Arm
Number analyzed (Participants) | 20
DSA Relative Intensity Score
  DSA RIS @ Transplant | 3.21 (2.86)
  DSA RIS @ Month 1 | 0.79 (1.69)
  DSA RIS @ Month 3 | 0.64 (1.97)
  DSA RIS @ Month 6: number analyzed (Participants) | 18
  DSA RIS @ Month 6 | 0.93 (2.70)
  DSA RIS @ Month 9: number analyzed (Participants) | 17
  DSA RIS @ Month 9 | 0.86 (2.26)
  DSA RIS @ Month 12: number analyzed (Participants) | 17
  DSA RIS @ Month 12 | 1.14 (2.49)

3. Secondary Outcome: Tolerability as Defined by the Number of Subjects Discontinuing the Study Medication
Description: To observe the tolerability as defined by the number of subjects discontinuing the study medication.
Time Frame: 12 months
Population: All participants enrolled were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus Extended-Release Arm
Number analyzed (Participants) | 20
Participants | 3

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events and severe adverse events were collected and reported in all enrolled participants who received study drug.
Arm/Group | Tacrolimus Extended-Release Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Extended-Release Arm (N=20)
Bacteremia (Blood and lymphatic system disorders) | 1
Diabetic ketoacidosis (DKA) (General disorders) | 1
Incisional abscess and acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Extended-Release Arm (N=20)
Mouth ulcer (Immune system disorders) | 1
Perinephric fluid collection (Renal and urinary disorders) | 1
BKAN Grade 2 with stable Serum Creatinine (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
Small sample size; Early withdrawal of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT03194321/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03194321/ICF_001.pdf